CLINICAL TRIAL: NCT03709199
Title: The Effect of Intensive Care Unit Therapies and Mechanical Ventilation Strategy on Long Term Outcome in Pediatric ARDS A Follow-up of the Real-time Effort Driven VENTilator Management Study (REDvent)
Brief Title: Long Term Follow up of Children Enrolled in the REDvent Study
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Robinder Khemani, Principal Investigator, Children's Hospital Los Angeles
Other Study IDs: CHLA-18-00354
Record Dates: First submitted 2018-08-30; First posted 2018-10-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Distress Syndrome, Adult; Ventilator-Induced Lung Injury; Neurocognitive Dysfunction; Quality of Life; Respiration Disorders
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury; Cognition Disorders; Respiration Disorders | interventions — Spirometry; Respiratory Function Tests; Functional Residual Capacity; Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ventilation Inhomogeneity — Ventilation inhomogeneity will be measured using the Lung Clearance Index (LCI), derived from multiple breath Nitrogen washout during tidal breathing, measured by a mouthpiece or mask covering nose and mouth.
  Other Names: Lung Clearance Index
Diagnostic Test: Diaphragm Ultrasound — Diaphragm thickness and contractile activity measured during tidal breathing.
Diagnostic Test: Respiratory Inductance Plethysmography — Measure of thoraco-abdominal asynchrony during tidal breathing
  Other Names: Phase Angle
Diagnostic Test: Spirometry — Measurement of Forced Expiratory Volume (FEV1), Forced Vital Capacity and other lung volumes using standard pulmonary function techniques
  Other Names: Pulmonary Function Tests
Diagnostic Test: Functional Residual Capacity — Measurement using body box plethysmography of functional residual capacity and other lung volumes using standard pulmonary function techniques
  Other Names: Pulmonary Function Tests
Diagnostic Test: MIP/MEP — Measurement of maximal inspiratory and expiratory pressures during airway occlusion
Diagnostic Test: 6 minute walk test — Measurement of cardio-respiratory function and capabilities during treadmill walking for 6 minutes.
Diagnostic Test: Neurocognitive Testing — Detailed in person neuro-cognitive testing using standardized inventories using either the Battelle Developmental Inventory, second edition (Battelle-2) (age birth to 5 years 11 months) and the Wechsler Intelligence Scale for Children, fifth edition (WISC-5, for age 6 years to 19 years).
Diagnostic Test: Emotional Health Assessment — In person and written assessments of children and parents using the Behavioral Assessment System for Children, third edition (BASC-3) for children ≥ 2 years and the UCLA PTSD Reaction Index (UCLA RI) for children ≥ 8 years.
Diagnostic Test: Health Related Quality of Life — Standardized instruments to assess (in person, over the phone, or via mail) health related quality of life in children. Parent and child questionnaires.
  Other Names: PEDS-QL
Diagnostic Test: Functional Status — Survey of overall functional status, administrated by asking a series of questions to patient and families.
  Other Names: Functional Status Scale
Diagnostic Test: Respiratory Status Questionnaire — Survey of respiratory health, administrated by asking a series of questions to patient and families.

SUMMARY:
This is a prospective observational follow-up study of children enrolled in a single center randomized controlled trial (REDvent).

Nearly 50% of adult Acute Respiratory Distress Syndrome (ARDS) survivors are left with significant abnormalities in pulmonary, physical, neurocognitive function and Health Related Quality of Life (HRQL) which may persist for years.Data in pediatric ARDS (PARDS) survivors is limited. More importantly, there are no data identifying potentially modifiable factors during ICU care which are associated with long term impairments, which may include medication choices, or complications from mechanical ventilator (MV) management in the ICU including ventilator induced lung injury (VILI) or ventilator induced diaphragm dysfunction (VIDD).

The Real-time effort driven ventilator (REDvent) trial is testing a ventialtor management algorithm which may prevent VIDD and VILI. VIDD and VILI have strong biologic plausibility to affect the post-ICU health of children with likely sustained effects on lung repair and muscle strength. Moreover, common medication choices (i.e. neuromuscular blockade, corticosteroids) or other complications in the ICU (i.e. delirium) are likely to have independent effects on the long term health of these children. This proposed study will obtain serial follow-up of subjects enrolled in REDvent (intervention and control patients). The central hypothesis is that preventing VIDD, VILI and shortening time on MV will have a measureable impact on longer term function by mitigating abnormalities in pulmonary function (PFTs), neurocognitive function and emotional health, functional status and HRQL after hospital discharge for children with PARDS.

For all domains, the investigators will determine the frequency, severity and trajectory of recovery of abnormalities amongst PARDS survivors after ICU discharge, identify risk factors for their development, and determine if they are prevented by REDvent. They will leverage the detailed and study specific respiratory physiology data being obtained in REDvent, and use a variety of multi-variable models for comprehensive analysis. Completion of this study will enable the investigators to identify ICU related therapies associated with poor long term outcome, and determine whether they can be mitigated by REDvent.

ELIGIBILITY:
Inclusion Criteria:

1. Children > 1 month (at least 44 weeks Corrected Gestational Age) and ≤ 18 years of age AND
2. Supported on mechanical ventilation for pulmonary parenchymal disease (i.e., pneumonia, bronchiolitis, Pediatric Acute Respiratory Distress Syndrome (PARDS)) with Oxygen Saturation Index (OSI) ≥ 5 or Oxygenation Index (OI) ≥4 115 AND
3. Who are within 48 hours of initiation of invasive mechanical ventilation (allow for up to 72 hours for those transferred from another institution) AND
4. Enrolled in the REDvent Study

Exclusion Criteria (1-5 are REDvent exclusion):

1. Contraindications to use of an esophageal catheter (i.e. severe mucosal bleeding, nasal encephalocele, transphenoidal surgery) OR
2. Contraindications to use of RIP bands (i.e. omphalocele, chest immobilizer or cast) OR
3. Conditions precluding diaphragm ultrasound measurement (i.e. abdominal wall defects, pregnancy) OR
4. Conditions precluding conventional methods of weaning (i.e., status asthmaticus, severe lower airway obstruction, critical airway, intracranial hypertension, Extra Corporeal Life Support (ECLS), intubation for UAO, tracheostomy, DNR, severe chronic respiratory failure, spinal cord injury above lumbar region, cyanotic heart disease (unrepaired or palliated)) OR
5. Primary Attending physician refuses (will be cleared with primary attending before approaching the patient) OR
6. Death in the ICU OR
7. New DNR orders during acute illness in ICU OR
8. Primary Language not English or Spanish OR
9. Children in foster care or a ward of the state.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a long term follow-up of children already enrolled in the RED-vent study.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation In-homogeneity using lung clearance index with nitrogen washout | 6 months after ICU discharge
  Measured by lung clearance index during multiple breath nitrogen washout testing reported as percent predicted based on age and height as well as a raw number typically ranging from 5-15.
Neurocognitive function using a standardized score derived from Batelle-2 or WISC-5 cognitive tests | 3 months after ICU discharge
  Standardized IQ-like score derived from Batelle-2 or WISC-5 cognitive tests based on age. Children < 6 years will receive the Batelle-2 and children >=6 will receive the WISC-5. Overall score will be use for analysis with a higher value indicating better cognitive function. The range of "average" cognitive function lies between 90-109. Both tests are scored on the same scale
Health Related Quality of Life as measured by PedsQL generic core scale | 3 months after ICU discharge
  PedsQL generic core scale, with range from 0-100, with the higher score indicating better health related quality of life
Functional Status as measured by the pediatric functional status scale | 3 months after ICU discharge
  Functional status scale which is scored from normal (score =1) to very severe dysfunction (score =5) in each of 6 domains. The sum score of all domains will be used for analysis, yielding a minimum possible score of 6 and a maximum possible score of 30. Analysis will focus on a change in FSS from baseline (assessed as functional status 1 month prior to ICU admission). An increase in the FSS from baseline to 3 months will be considered as a decline in functional status.

SECONDARY OUTCOMES:
Functional Residual Capacity (Lung volume at end-expiration). | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Measured by body box plethysmography and nitrogen washout techniques, normalized by age, height and gender. Values below or above normative values will be considered abnormal.
Functional Residual Capacity (Lung volume at end-expiration). | 6 months after ICU discharge
  Measured by body box plethysmography and nitrogen washout techniques, normalized by age, height and gender. Values below or above normative values will be considered abnormal.
Phase Angle (a measure of thoraco-abdominal asynchrony and abnormal respiratory mechanics) | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Respiratory Inductance Plethysmography belts are used during tidal breathing to measure thoraco-abdominal asyncrhony. Higher values will be considered abnormal with a range from 0-180.
Phase Angle (a measure of thoraco-abdominal asynchrony and abnormal respiratory mechanics) | 6 Months after ICU Discharge
  Respiratory Inductance Plethysmography belts are used during tidal breathing to measure thoraco-abdominal asyncrhony. Higher values will be considered abnormal with a range from 0-180.
Diaphragm Thickness on exhalation | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Diaphragm ultrasound measurement of thickness at end exhalation measured in zone of apposition of right hemi-diaphragm
Diaphragm Thickness on exhalation | 6 months after ICU discharge
  Diaphragm ultrasound measurement of thickness at end exhalation measured in zone of apposition of right hemi-diaphragm
Diaphragm Thickness on inspiration | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Diaphragm ultrasound measurement of thickness at end inspiration measured in zone of apposition of right hemi-diaphragm
Diaphragm Thickness on inspiration | 6 months after ICU discharge
  Diaphragm ultrasound measurement of thickness at end inspiration measured in zone of apposition of right hemi-diaphragm
Diaphragm Thickening fraction (measure of contractile activity) | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Diaphragm ultrasound measurement calculated as (thickness at end inspiration-thickness at end expiration)/(thickness at end expiration) measured in zone of apposition of right hemi-diaphragm.
Diaphragm Thickening fraction (measure of contractile activity) | 6 months after ICU discharge
  Diaphragm ultrasound measurement calculated as (thickness at end inspiration-thickness at end expiration)/(thickness at end expiration) measured in zone of apposition of right hemi-diaphragm.
Ventilation In-homogeneity using lung clearance index with nitrogen washout | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Measured by lung clearance index during multiple breath nitrogen washout testing reported as percent predicted based on age and height as well as a raw number typically ranging from 5-15.
Forced Expiratory Volume in 1 second (FEV1) | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Spirometry based measures of pulmonary function of forced expiratory volume, normalized based on age, height, and gender and reported as percent predicted.
Forced Expiratory Volume in 1 second (FEV1) | 6 months after ICU discharge
  Spirometry based measures of pulmonary function of forced expiratory volume, normalized based on age, height, and gender and reported as percent predicted.
Forced Vital Capacity (FVC) | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Spirometry based measures of pulmonary function of forced vital capacity, normalized based on age, height, and gender and reported as percent predicted.
Forced Vital Capacity (FVC) | 6 months after ICU discharge
  Spirometry based measures of pulmonary function of forced vital capacity, normalized based on age, height, and gender and reported as percent predicted.
Forced expiratory flow at 25-75% (FEF 25-75) | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Spirometry based measures of pulmonary function of forced expiratory flow at 25-75% of breath, normalized based on age, height, and gender and reported as percent predicted.
Forced expiratory flow at 25-75% (FEF 25-75) | 6 months post ICU discharge
  Spirometry based measures of pulmonary function of forced expiratory flow at 25-75% of breath, normalized based on age, height, and gender and reported as percent predicted.
VT - tidal volume from spirometry during tidal breathing | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Lung volume measurements obtained during tidal breathing, normalized in ml/kg ideal body weight.
VT - tidal volume from spirometry during tidal breathing | 6 months after ICU discharge
  Lung volume measurements obtained during tidal breathing, normalized in ml/kg ideal body weight.
Total Lung Capacity- TLC measured during spirometry | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Lung volume measurements obtained during pulmonary function tests with spirometry and body box plethysmography to calculate total lung capacity, normalized by age, height and gender.
Total Lung Capacity- TLC measured during spirometry | 6 months after ICU discharge
  Lung volume measurements obtained during pulmonary function tests with spirometry and body box plethysmography to calculate total lung capacity, normalized by age, height and gender.
Forced vital capacity- measured during spirometry | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Lung volume measurements obtained during pulmonary function tests with spirometry to calculate forced vital capacity, normalized by age, height and gender.
Forced vital capacity- measured during spirometry | 6 months after ICU discharge
  Lung volume measurements obtained during pulmonary function tests with spirometry to calculate forced vital capacity, normalized by age, height and gender.
Respiratory Muscle Strength Maximum inspiratory pressure (MIP) | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Maximal inspiratory pressure measurements during airway occlusion in cm H20
Respiratory Muscle Strength Maximum inspiratory pressure (MIP) | 6 months after ICU discharge
  Maximal inspiratory pressure measurements during airway occlusion in cm H20
Respiratory Muscle Strength Maximum expiratory pressure (MEP) | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Maximal expiratory pressure measurements during airway occlusion in cm H20
Respiratory Muscle Strength Maximum expiratory pressure (MEP) | 6 months after ICU discharge
  Maximal expiratory pressure measurements during airway occlusion in cm H20
Neurocognitive function using a standardized score derived from Batelle-2 or WISC-5 cognitive tests | 12 months after ICU discharge
  Standardized IQ-like score derived from Batelle-2 or WISC-5 cognitive tests. Overall score will be use for analysis with a higher value indicating better cognitive function. The range of "average" cognitive function lies between 90-109.
Health Related Quality of Life as measured by PedsQL generic core scale | ICU discharge
  PedsQL generic core scale, with range from 0-100, with the higher score indicating better health related quality of life
Health Related Quality of Life as measured by PedsQL generic core scale | 1 month after ICU discharge
  PedsQL generic core scale, with range from 0-100, with the higher score indicating better health related quality of life
Health Related Quality of Life as measured by PedsQL generic core scale | 2 months after ICU discharge
  PedsQL generic core scale, with range from 0-100, with the higher score indicating better health related quality of life
Health Related Quality of Life as measured by PedsQL generic core scale | 6 months after ICU discharge
  PedsQL generic core scale, with range from 0-100, with the higher score indicating better health related quality of life
Health Related Quality of Life as measured by PedsQL generic core scale | 12 months after ICU discharge
  PedsQL generic core scale, with range from 0-100, with the higher score indicating better health related quality of life
Functional Status as measured by the pediatric functional status scale | ICU discharge
  Functional status scale which is scored from normal (score =1) to very severe dysfunction (score =5) in each of 6 domains. The sum score of all domains will be used for analysis, yielding a minimum possible score of 6 and a maximum possible score of 30. Analysis will focus on a change in FSS from baseline (assessed as functional status 1 month prior to ICU admission). An increase in the FSS from baseline will be considered as a decline in functional status.
Functional Status as measured by the pediatric functional status scale | 1 month after ICU discharge
  Functional status scale which is scored from normal (score =1) to very severe dysfunction (score =5) in each of 6 domains. The sum score of all domains will be used for analysis, yielding a minimum possible score of 6 and a maximum possible score of 30. Analysis will focus on a change in FSS from baseline (assessed as functional status 1 month prior to ICU admission). An increase in the FSS from baseline will be considered as a decline in functional status.
Functional Status as measured by the pediatric functional status scale | 2 months after ICU discharge
  Functional status scale which is scored from normal (score =1) to very severe dysfunction (score =5) in each of 6 domains. The sum score of all domains will be used for analysis, yielding a minimum possible score of 6 and a maximum possible score of 30. Analysis will focus on a change in FSS from baseline (assessed as functional status 1 month prior to ICU admission). An increase in the FSS from baseline will be considered as a decline in functional status.
Functional Status as measured by the pediatric functional status scale | 6 months after ICU discharge
  Functional status scale which is scored from normal (score =1) to very severe dysfunction (score =5) in each of 6 domains. The sum score of all domains will be used for analysis, yielding a minimum possible score of 6 and a maximum possible score of 30. Analysis will focus on a change in FSS from baseline (assessed as functional status 1 month prior to ICU admission). An increase in the FSS from baseline will be considered as a decline in functional status.
Functional Status as measured by the pediatric functional status scale | 12 months after ICU discharge
  Functional status scale which is scored from normal (score =1) to very severe dysfunction (score =5) in each of 6 domains. The sum score of all domains will be used for analysis, yielding a minimum possible score of 6 and a maximum possible score of 30. Analysis will focus on a change in FSS from baseline (assessed as functional status 1 month prior to ICU admission). An increase in the FSS from baseline will be considered as a decline in functional status.
Respiratory Status - questionnaire detailing respiratory medications and therapies as well as healthcare utilization. | ICU discharge
  Series of questions to detail respiratory based morbidity
Respiratory Status - questionnaire detailing respiratory medications and therapies as well as healthcare utilization. | 1 month after ICU discharge
  Series of questions to detail respiratory based morbidity
Respiratory Status - questionnaire detailing respiratory medications and therapies as well as healthcare utilization. | 2 months after ICU discharge
  Series of questions to detail respiratory based morbidity
Respiratory Status - questionnaire detailing respiratory medications and therapies as well as healthcare utilization. | 3 months after ICU discharge
  Series of questions to detail respiratory based morbidity
Respiratory Status - questionnaire detailing respiratory medications and therapies as well as healthcare utilization. | 6 months after ICU discharge
  Series of questions to detail respiratory based morbidity
Respiratory Status - questionnaire detailing respiratory medications and therapies as well as healthcare utilization. | 12 months after ICU discharge
  Series of questions to detail respiratory based morbidity
Emotional Health Outcomes using the (BASC-3) to assess emotional and behavioral abnormalities and UCLA Reaction Index to assess post traumatic stress | 3 months after ICU discharge
  The Behavioral Assessment System for Children, third edition (BASC-3) for children ≥ 2 years will be used to assess for emotional and behavioral abnormalities as a survey tool. The UCLA PTSD Reaction Index (UCLA RI) will be used for children ≥ 8 years. The UCLA RI is a semi-structured interview assessing for exposure to traumatic events and PTS in children.
Emotional Health Outcomes using the (BASC-3) to assess emotional and behavioral abnormalities and UCLA Reaction Index to assess post traumatic stress | 12 months after ICU discharge
  The Behavioral Assessment System for Children, third edition (BASC-3) for children ≥ 2 years will be used to assess for emotional and behavioral abnormalities as a survey tool. The UCLA PTSD Reaction Index (UCLA RI) will be used for children ≥ 8 years. The UCLA RI is a semi-structured interview assessing for exposure to traumatic events and PTS in children.

OTHER OUTCOMES:
6 minute walk test | Prior to Hospital Discharge and no more than 1 month after ICU discharge
  Measure of cardio-respiratory function after treadmill walking
6 minute walk test | 6 months after ICU discharge
  Measure of cardio-respiratory function after treadmill walking

CONTACTS AND LOCATIONS:
Overall Officials: Robinder Khemani, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers